CLINICAL TRIAL: NCT01359995
Title: Topical Ganciclovir in Patients Receiving Penetrating Keratoplasty With Cytomegalovirus Endotheliitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: I-Jong Wang, Department of Ophthalmology
Other Study IDs: 201010033R
Record Dates: First submitted 2011-05-16; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Cytomegalovirus Endotheliitis
Keywords: cytomegalovirus endotheliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to evaluate the outcomes of topical ganciclovir in patients with cytomegalovirus endotheliitis receiving penetrating keratoplasty at National Taiwan University hospital.

DETAILED DESCRIPTION:
In this study, we recruit 7 immunocompetent patients with unexplained graft failures, which mimicked herpetic anterior uveitis and graft rejection initially, were diagnosed as CMV endotheliitis after aqueous tapping for CMV polymerase chain reaction (PCR). Topical ganciclovir was used to control and prevent the reactivation of CMV without systemic application and their clinical courses were presented after this treatment modality.

The purpose of this study was to evaluate the outcomes of topical ganciclovir in patients with cytomegalovirus endotheliitis receiving penetrating keratoplasty at National Taiwan University hospital.

ELIGIBILITY:
Inclusion Criteria:

* immunocompetent patients with positive results of the CMV PCR (polymerase chain reaction) from aqueous humor tapping receiving penetrating keratoplasty

Exclusion Criteria:

* patients receiving systemic or intravitreal ganciclovir before topical ganciclovir use

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4 men, 3 women, aged 40-90 years old
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
clinical courses before and after topical ganciclovir in patients with CMV endotheliitis | participants will be monitored after receiving topical ganciclovir,an expected average of 1 year
  evaluations including aqueous PCR for CMV, endothelium cell density on confocal microscopy,degree of anterior chamber inflammation..

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, M.D. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Koizumi N, Suzuki T, Uno T, Chihara H, Shiraishi A, Hara Y, Inatomi T, Sotozono C, Kawasaki S, Yamasaki K, Mochida C, Ohashi Y, Kinoshita S. Cytomegalovirus as an etiologic factor in corneal endotheliitis. Ophthalmology. 2008 Feb;115(2):292-297.e3. doi: 10.1016/j.ophtha.2007.04.053. Epub 2007 Jul 31. PMID 17669498
- [Background] Chee SP, Bacsal K, Jap A, Se-Thoe SY, Cheng CL, Tan BH. Clinical features of cytomegalovirus anterior uveitis in immunocompetent patients. Am J Ophthalmol. 2008 May;145(5):834-40. doi: 10.1016/j.ajo.2007.12.015. Epub 2008 Feb 6. PMID 18255045
- [Background] Anshu A, Chee SP, Mehta JS, Tan DT. Cytomegalovirus endotheliitis in Descemet's stripping endothelial keratoplasty. Ophthalmology. 2009 Apr;116(4):624-30. doi: 10.1016/j.ophtha.2008.10.031. Epub 2009 Feb 4. PMID 19195708